CLINICAL TRIAL: NCT05678751
Title: Establishment of a Rapid Detection Method for Microorganisms in the Lower Genital Tract Using MALDI-TOF MS and Its Clinical Application in Infertility
Brief Title: Rapid Detection Method for Microorganisms in the Lower Genital Tract
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: yzy_00159
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-07

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vaginal and cervical secretions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: patients with infertility
  Interventions: Diagnostic Test: lower genital tract microorganisms detection using Matrix-Assisted Laser Desorption/Ionization Time of Flight Mass Spectrometry (MALDI-TOF MS)
- control group: women that are capable of spontaneous intrauterine pregnanc
  Interventions: Diagnostic Test: lower genital tract microorganisms detection using Matrix-Assisted Laser Desorption/Ionization Time of Flight Mass Spectrometry (MALDI-TOF MS)

INTERVENTIONS:
Diagnostic Test: lower genital tract microorganisms detection using Matrix-Assisted Laser Desorption/Ionization Time of Flight Mass Spectrometry (MALDI-TOF MS) — Detection of pathogens and microorganisms in the lower genital tract of infertile and spontaneously pregnant women by a new MALDI-TOF MS-based technique

SUMMARY:
Mycoplasma, chlamydia, and gonococcal infection of the female lower genital tract can lead to infertility and various adverse pregnancy outcomes. The lower genital tract bacterial community status type (CST) is closely related to genital tract infection and reproductive health. However, there is a need for a rapid, accurate, stable, and economical detection method to detect the above pathogens and CST at the same time, so there is also a need for evaluation of the correlation between each pathogen infection and CST. Matrix assisted laser desorption ionization time-of-flight mass spectrometry (MALDI-TOF MS) is more stable and accurate than traditional detection methods such as culture and staining. It can simultaneously detect a variety of microorganisms and their subtypes, while the high-throughput sequencing method is faster and more economical, which is suitable for detecting multiple microorganisms in clinical practice. The research group has established a perfect MALDI-TOF MS platform in the early stage and put it into clinical testing. This project will establish a new rapid detection method for lower genital tract microorganisms based on MALDI-TOF MS. Then, examine the lower genital tract microecology of infertile patients and healthy women using the newly developed method. At last, analyze the correlation between pathogen infection, CST status, and infertility. This project will solve the practical work needs of clinicians for a comprehensive assessment of female lower genital tract CST and common pathogen infection and fill in the technical gaps in the microbial examination of the lower genital tract.

ELIGIBILITY:
Inclusion Criteria:

Case group:

1) Female aged 18-40 2) Regular menstrual cycle 2) Conform to the clinical diagnosis of infertility 3) No sexual life 3 days before the examination control group:

1. Female aged 18-40
2. Regular menstrual cycle
3. Patients who did pre-pregnancy consultation in our hospital, pregnant at the time of 3-month follow-up
4. No sexual life 3 days before the examination -

Exclusion Criteria:

Case group:

1. Infertility due to malformation of reproductive tract
2. Infertility caused by endocrine factors such as polycystic ovary syndrome, premature ovarian failure and severe hyperthyroidism
3. Infertility due to male factors
4. Patients with malignant tumors
5. Patients with autoimmune diseases
6. Patients with severe heart, kidney and other basic diseases
7. Patients who consumed antibiotics 3 days before the examination
8. Have the habit of smoking and drinking

Control group:

1. Pregnancy by various assisted reproductive means
2. Patients with malignant tumors
3. Patients with autoimmune diseases
4. Patients with severe heart, kidney and other basic diseases
5. Patients who consumed antibiotics 3 days before the examination
6. Have the habit of smoking and drinking

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The target disease of this study is infertility, so its not based on self-representation of gender identity
Study Population: Women of childbearing age who can spontaneous pregnancy and infertile women
Sampling Method: Non-Probability Sample
Enrollment: 228 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Lower genital tract pathogen | at recruitment
  Ureaplasma urealyticum, mycoplasma hominis, chlamydia antigen, gonococcus
Lower genital CST | at recruitment
  Lactobacillus crispatus, Lactobacillus gasseri, Lactobacillus iners, Lactobacillus jensenii

CONTACTS AND LOCATIONS:
Overall Officials: Zhiying Yu, M.D., Study Chair — Shenzhen Second People's Hospital; Wenlan Liu, PhD, Study Director — Shenzhen Second People's Hospital

IPD SHARING:
Plan to Share IPD: Undecided
Because this study involves private information related to patient reproduction, we may not fully disclose subject details, but we will evaluate applicants and give non-private data by email, etc., when necessary.

REFERENCES:
- [Background] Chen YJ, Hsu TF, Huang BS, Tsai HW, Chang YH, Wang PH. Postoperative maintenance levonorgestrel-releasing intrauterine system and endometrioma recurrence: a randomized controlled study. Am J Obstet Gynecol. 2017 Jun;216(6):582.e1-582.e9. doi: 10.1016/j.ajog.2017.02.008. Epub 2017 Feb 15. PMID 28209488
- [Background] Carey AJ, Beagley KW. Chlamydia trachomatis, a hidden epidemic: effects on female reproduction and options for treatment. Am J Reprod Immunol. 2010 Jun;63(6):576-86. doi: 10.1111/j.1600-0897.2010.00819.x. Epub 2010 Feb 28. PMID 20192953
- [Background] Chee WJY, Chew SY, Than LTL. Vaginal microbiota and the potential of Lactobacillus derivatives in maintaining vaginal health. Microb Cell Fact. 2020 Nov 7;19(1):203. doi: 10.1186/s12934-020-01464-4. PMID 33160356
- [Background] Smith SB, Ravel J. The vaginal microbiota, host defence and reproductive physiology. J Physiol. 2017 Jan 15;595(2):451-463. doi: 10.1113/JP271694. Epub 2016 May 5. PMID 27373840
- [Background] Dunlop AL, Satten GA, Hu YJ, Knight AK, Hill CC, Wright ML, Smith AK, Read TD, Pearce BD, Corwin EJ. Vaginal Microbiome Composition in Early Pregnancy and Risk of Spontaneous Preterm and Early Term Birth Among African American Women. Front Cell Infect Microbiol. 2021 Apr 29;11:641005. doi: 10.3389/fcimb.2021.641005. eCollection 2021. PMID 33996627

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT05678751/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/51/NCT05678751/ICF_001.pdf